CLINICAL TRIAL: NCT04969016
Title: A Prospective Randomized Controlled Trial Comparing Cyanoacrylate Skin Adhesive With Staple for Surgical Incision Closure After Laparoscopic / Robotic Bowel Resection
Brief Title: A Study Comparing Skin Adhesive With Staple for Surgical Incision Closure After Laparoscopic / Robotic Bowel Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-1023
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Benign or Malignant Diseases With Indication for Laparoscopic or Robotic Colorectal Resection
MeSH Terms: interventions — Surgical Staplers

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSA (liquid skin adhesive) (Experimental): surgical wound closure with liquid skin adhesive (LiquiBand®)
  Interventions: Procedure: LSA (liquid skin adhesive)
- Stapler (Active Comparator): surgical wound closure with stapler
  Interventions: Procedure: stapler

INTERVENTIONS:
Procedure: LSA (liquid skin adhesive) — surgical wound closure with liquid skin adhesive (LiquiBand®)
  Arms: LSA (liquid skin adhesive)
Procedure: stapler — surgical wound closure with stapler
  Arms: Stapler

SUMMARY:
INTRODUCTION

Liquid skin adhesive (LSA) has benefits over other closure methods. Especially it is less invasive, quicker to apply, and better in cosmesis. Also LSA applied wounds need no post-care and its water-proof nature allows patients to take a shower immediate postoperative periods. While traditional sutures and skin staples are invasive and have infection chance requiring regular wound dressings, LSA is resistant against both water and microbial infection without need for postoperative dressings. Thus LSA-applied wounds need no professional care saving wound management cost.

This study investigated not only the safety and efficacy of LSA, but also the cost-effectiveness in the context of total wound management resources including man-power, time, and cost.

STUDY OBJECTIVE

Primary end point of this study is time requiring to manage surgical wound calculated as man hour. Secondary end points are wound related complication and cost for management of surgical wound.

STATISTICAL ANALYSIS

The target number of the enrollment were calculated under the hypothesis that the wound management time for stapler group would be 1560 sec and that for LSA group be 264 sec with 10% drop-out rate. The sample number calculation formula of the t-test for independent 2 groups were used. For two-sided validation with the significance level of 0.05, and the power of 0.8, 29 patients for each group were estimated.

DETAILED DESCRIPTION:
STUDY DESIGN

1. Screening: replaced with preoperative examination

   * chest X-ray, CBC, CEA, BUN/Cr, OT/PT, glucose, EKG, abdominopelvic CT (optional), chest CT (optional), PET-CT(optional), MRI(optional)
2. Subject

   * Experimental group: surgical wound closure with liquid skin adhesive
   * Control group: surgical wound closure with stapler
3. Randomization The patients were randomized just before surgery after anesthesia and were randomly assigned to either experimental or control group as to computer-generated random number in 1:1 manner.
4. Study schedule

   * The enrolled patients received an elective surgery within 30 days after screening.
   * Surgical wound managers checked every enrolled patient from immediate postoperative period until discharge at least 1 time per day. Surgical wound managers were either surgical hospitalists (general surgery boards), surgical residents, or wound care specialist nurses. Incompletely healed wounds until discharge were managed regularly in out-patient clinics additionally. If wound complications were noted at any time point, standard treatment was given according to the patient's status regardless of assigned groups
5. Wound management

   * Wound healing time was defined as the time period from the moment of skin closure to the point when a surgical wound manager declared that the wound was healed either during admission or in out-patient clinic. For LSA group, wound closure time was measured in second starting from when LiquiBand® was applied to the first skin incision to when LiquiBand® was completely dried up in all skin incisions. For stapler group, it was measured as the whole time in second spent to apply skin staplers to all skin incisions in about 1cm interval without any dehiscence.
   * Surgical wound management was performed at least once a day in all patients. Wound management time was measured when surgical wound manager inspected and performed wound dressing as required. It was defined as time in second starting from the moment a patient completely took off tops to the moment a surgical wound manager took off gloves on the completion of dressing.
   * The complete wound healing was declared by surgical wound managers for wounds that have injections less than 2mm, no skin color change on the edges, no dehiscence on the inspection under white light.
   * Wound management time and cost were analyzed separately for event places (during admission - and out-patient clinic). Wound management time was compensated as to surgical wound managers and converted in to man-hour. The compensation constant was defined to reduce bias by performer assuming the skill level of wound management was different among surgical wound managers. The surgical hospitalists who were general surgery boards were found to be the most skillful, therefore the constant for them was defined as 1. The constants for surgical residents and wound care specialist nurses were defined as 0.6 and 0.8 respectively.
   * The total wound management cost included dressing fee and material cost. Generally, for normal wounds, adhesive foam dressings were used and for complicated wounds, gauzes and vicryl sutures were used as necessary. In Korean National Insurance System, dressing material costs were classified as the benefit service charge which was reimbursed by National Health Insurance Cooperation (NHIC) and the non-benefit service charge which a patient should pay all. Every dressing material was check whether the benefit service or the non-benefit service and the cost was recorded accordingly.

ELIGIBILITY:
Inclusion Criteria:

A. 19-year-old or older adults B. elective laparoscopic or robotic colorectal resection C. clean-contaminated surgery without any intraoperative contamination D. The longest incision should be 15cm or shorter E. participant should voluntarily sign inform consent form

Exclusion Criteria:

A. emergency surgery or conversion-to-open surgery B. the longest skin incision longer than 15cm C. intraoperative contamination due to intestinal perforation or any other reason D. ECOG grade 3 or higher E. patients who are not be able to receive surgery within 30 days after screening F. patients who are refused to sign the informed consent form voluntarily

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-10-22 (Estimated); Study Completion 2021-10-22 (Estimated)

PRIMARY OUTCOMES:
Total management time of surgical wound | postoperative day 60
  Wound management time was defined as the time period from the moment of skin closure to the point when the wound was healed either during admission or in out-patient clinic. For LSA group, skin closure time was measured in second starting from when LiquiBand® was applied to the first skin incision to when LiquiBand® was completely dried up in all skin incisions. For stapler group, it was measured as the whole time in second spent to apply skin staplers to all skin incisions in about 1cm interval.
  Wound management was performed at least once a day in all patients. Time was measured when surgical wound manager inspected and performed wound dressing as required. It was defined as time in second starting from the moment a patient completely took off tops to the moment a surgical wound manager took off gloves on the completion of dressing.

SECONDARY OUTCOMES:
Surgical wound related complication | postoperative day 60
  Surgical wound related complication is classified as erythema, edema, tenderness, inflammation, discharge, surgical site infection and dehiscence.
Total management costs of surgical wound | postoperative day 60
  The total wound management cost included dressing fee and material cost. Generally, for normal wounds, adhesive foam dressings were used and for complicated wounds, gauzes and vicryl sutures were used as necessary. In Korean National Insurance System, dressing material costs were classified as the benefit service charge which was reimbursed by National Health Insurance Cooperation (NHIC) and the non-benefit service charge which a patient should pay all. Every dressing material was check whether the benefit service or the non-benefit service and the cost was recorded accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Byung Soh Min, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jan H, Waters N, Haines P, Kent A. LiquiBand(R) Surgical S topical adhesive versus sutures for the closure of laparoscopic wounds. A randomized controlled trial. Gynecol Surg. 2013;10(4):247-252. doi: 10.1007/s10397-013-0805-5. Epub 2013 Jul 10. PMID 24273476
- [Background] Dowson CC, Gilliam AD, Speake WJ, Lobo DN, Beckingham IJ. A prospective, randomized controlled trial comparing n-butyl cyanoacrylate tissue adhesive (LiquiBand) with sutures for skin closure after laparoscopic general surgical procedures. Surg Laparosc Endosc Percutan Tech. 2006 Jun;16(3):146-50. doi: 10.1097/00129689-200606000-00005. PMID 16804456
- [Background] Koonce SL, Eck DL, Shaddix KK, Perdikis G. A prospective randomized controlled trial comparing N-butyl-2 cyanoacrylate (Histoacryl), octyl cyanoacrylate (Dermabond), and subcuticular suture for closure of surgical incisions. Ann Plast Surg. 2015 Jan;74(1):107-10. doi: 10.1097/SAP.0b013e318289856f. PMID 24905134
- [Background] Fraeman KH, Reynolds MW, Vaughn BB, Hart JC. Patient outcomes associated with 2-octyl cyanoacrylate topical skin adhesive in coronary artery bypass graft surgery. Surg Infect (Larchmt). 2011 Aug;12(4):307-16. doi: 10.1089/sur.2010.062. PMID 21859334
- [Background] Bartenstein DW, Cummins DL, Rogers GS. A Prospective, Randomized, Single-Blind Study Comparing Cyanoacrylate Adhesives to Sutures for Wound Closure in Skin Cancer Patients. Dermatol Surg. 2017 Nov;43(11):1371-1378. doi: 10.1097/DSS.0000000000001200. PMID 28595249
- [Background] Malhotra V, Dayashankara Rao JK, Arya V, Sharma S, Singh S, Luthra P. Evaluating the use of octyl-2-cyanoacrylate in unilateral cleft lip repair. Natl J Maxillofac Surg. 2016 Jul-Dec;7(2):153-158. doi: 10.4103/0975-5950.201364. PMID 28356686
- [Background] Martin JG, Hollenbeck ST, Janas G, Makar RA, Pabon-Ramos WM, Suhocki PV, Miller MJ, Sopko DR, Smith TP, Kim CY. Randomized Controlled Trial of Octyl Cyanoacrylate Skin Adhesive versus Subcuticular Suture for Skin Closure after Implantable Venous Port Placement. J Vasc Interv Radiol. 2017 Jan;28(1):111-116. doi: 10.1016/j.jvir.2016.08.009. Epub 2016 Nov 9. PMID 27836404
- [Background] Chen CT, Choi CL, Suen DT, Kwong A. A prospective randomised controlled trial of octylcyanoacrylate tissue adhesive and standard suture for wound closure following breast surgery. Hong Kong Med J. 2016 Jun;22(3):216-22. doi: 10.12809/hkmj154513. Epub 2016 Apr 22. PMID 27101789
- [Background] Buchweitz O, Frye C, Moeller CP, Nugent W, Krueger E, Nugent A, Biel P, Juergens S. Cosmetic outcome of skin adhesives versus transcutaneous sutures in laparoscopic port-site wounds: a prospective randomized controlled trial. Surg Endosc. 2016 Jun;30(6):2326-31. doi: 10.1007/s00464-015-4474-5. Epub 2015 Oct 1. PMID 26428200
- [Background] Van Haute C, Tailly T, Klockaerts K, Ringoir Y. Sutureless circumcision using 2-Octyl cyanoacrylate results in more rapid and less painful procedures with excellent cosmetic satisfaction. J Pediatr Urol. 2015 Jun;11(3):147.e1-5. doi: 10.1016/j.jpurol.2015.02.013. Epub 2015 Mar 20. PMID 25910797
- [Background] Imbuldeniya AM, Rashid A, Murphy JP. A comparison of 2-octyl cyanoacrylate with nylon for wound closure of knee arthroscopy portals. J Wound Care. 2014 Sep;23(9):456-8, 460. doi: 10.12968/jowc.2014.23.9.456. PMID 25284299
- [Background] Ando M, Tamaki T, Yoshida M, Sasaki S, Toge Y, Matsumoto T, Maio K, Sakata R, Fukui D, Kanno S, Nakagawa Y, Yamada H. Surgical site infection in spinal surgery: a comparative study between 2-octyl-cyanoacrylate and staples for wound closure. Eur Spine J. 2014 Apr;23(4):854-62. doi: 10.1007/s00586-014-3202-5. Epub 2014 Feb 1. PMID 24487558
- [Background] Mudd CD, Boudreau JA, Moed BR. A prospective randomized comparison of two skin closure techniques in acetabular fracture surgery. J Orthop Traumatol. 2014 Sep;15(3):189-94. doi: 10.1007/s10195-013-0282-7. Epub 2013 Dec 31. PMID 24379118
- [Background] Soni A, Narula R, Kumar A, Parmar M, Sahore M, Chandel M. Comparing cyanoacrylate tissue adhesive and conventional subcuticular skin sutures for maxillofacial incisions--a prospective randomized trial considering closure time, wound morbidity, and cosmetic outcome. J Oral Maxillofac Surg. 2013 Dec;71(12):2152.e1-8. doi: 10.1016/j.joms.2013.08.029. PMID 24237777
- [Background] Julious SA, Owen RJ. A comparison of methods for sample size estimation for non-inferiority studies with binary outcomes. Stat Methods Med Res. 2011 Dec;20(6):595-612. doi: 10.1177/0962280210378945. Epub 2010 Oct 1. PMID 20889572